CLINICAL TRIAL: NCT05030688
Title: Comparison of the Effect of Ultrasound-guided Fascia Iliaca Compartment Block and PENG Block on Postoperative Analgesia Management in Patients Undergoing Hip Arthroplasty: A Multicentric, Randomized, Prospective Study.
Brief Title: Fascia Iliaca Compartment Block and PENG Block for Hip Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participant
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 20
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Hip Fractures; Hip Injuries; Hip Arthropathy
Keywords: Hip arthroplasty; Fascia iliaca compartment block; PENG block; Postoperative analgesia
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is fascia iliaca compartment block (FICB). The second one is PENG block group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient, and the outcomes assessor who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group FICB = Fascia iliaca compartment block (Active Comparator): FICB will be performed with a suprainguinal approach under US guidance. The probe will be placed sagittally to view the ilium and iliacus muscle. The probe will be moved medially and inferiorly along the inguinal ligament to view the femoral artery. The probe will then be moved superiorly and laterally along the inguinal ligament towards the anterior superior iliac crest to reach the lateral aspect of the femoral nerve. The deep circumflex artery will be visualized 1-2 cm cephalad to the inguinal ligament and superficial to the iliac fascia. The needle will be inserted with in-plane method 2-4 cm caudal to the inguinal ligament to reach below the fascia ilica. After the block site is confirmed with 5 ml of saline, 30 ml of local anesthetic solution containing 0.25% bupivacaine will be injected.
  Interventions: Other: Postoperative analgesia management
- Group PENG (Active Comparator): The probe will be placed on the anterior inferior iliac crest in the transverse plane. Then, the pubic ramus will be visualized by rotating 45 degrees. The femoral artery, iliopubic process and psoas muscle will be visualized. The needle will be punctured with the in-plane method to reach between the pubic ramus and the psoas tendon. After the block site is confirmed with 5 ml of saline, 30 ml of local anesthetic solution containing 0.25% bupivacaine will be injected.
  Interventions: Other: Postoperative analgesia management

INTERVENTIONS:
Other: Postoperative analgesia management — Intravenous 0.5 mg/kg tramodol and 400 mg ibuprofen will be administered to all patients 30 minutes before the end of the surgical procedure. In the postoperative period, patients will be administered ibuprofen iv 400 mg 3x1. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic.

SUMMARY:
Hip arthroplasty is one of the most common orthopedic procedures especially in elderly patients due to deformation of joint. Patients may complain severe pain due to the surgical trauma and the prosthesis. Regional anesthesia methods may be performed to reduce opioid consumption and opioid-related side effects. The hip joint consists of the femoral head and the acetabulum. Sensory innervation of the hip joint is provided by the femoral nerve, obturator nerve, articular branches of the sciatic nerve, and superior gluteal nerve. Because of the increasing use of ultrasound (US) in anesthesia practice, US-guided nerve blocks are widely used. One of the most used methods in the management of analgesia after hip surgery is the fascia iliaca compartment block (FICB). Pericapsular nerve group block (PENG block) is a novel fascial block defined by Arango et al. In this block, it is aimed to block the femoral nerve and the accessory obturatory nerve by injecting local anesthetic between the pubic ramus and the psoas tendon. This prospective, multicenter study aimed to compare the efficacy of PENG block and FICB for postoperative analgesia management in patients undergoing hip arthroplasty with a prosthesis. Our primary aim is to compare global recovery scores, and our secondary aim is to evaluate postoperative opioid consumption, pain scores (Numerical Rating Scale-NRS), and side effects (allergic reaction, nausea, vomiting, etc.) related with opioid use.

DETAILED DESCRIPTION:
Hip arthroplasty is one of the most common orthopedic procedures especially in elderly patients due to deformation of joint. Patients may complain severe pain due to the surgical trauma and the prosthesis. Opioid agents are commonly used for analgesia management. However, opioids have adverse effects such as nausea, vomiting, sedation and respiratory depression. Regional anesthesia methods may be performed to reduce opioid consumption and opioid-related side effects. The hip joint consists of the femoral head and the acetabulum. Sensory innervation of the hip joint is provided by the femoral nerve, obturator nerve, articular branches of the sciatic nerve, and superior gluteal nerve. Skin innervation of the lateral femur is provided by the lateral cutaneous femoral nerve. The upper anterior part of the thigh is innervated by the genitofemoral and ilioinguinal nerves. These nerves originate from the lumbar and sacral plexus. The innervation of the hip joint is complex, and the selection of the blocking technique is important after these operations.

Because of the increasing use of ultrasound (US) in anesthesia practice, US-guided nerve blocks are widely used. One of the most used methods in the management of analgesia after hip surgery is the fascia iliaca compartment block (FICB). FICB was first described in 1989 by Dalens et al. defined by. It is a popular regional anesthetic technique for surgical procedures involving the hip joint and femur. Since the local anesthetic agent is injected proximally under the fascia ilica, FICB can be considered as the anterior approach of the lumbar plexus blockade. It blocks the femoral nerve, obturator nerve, and lateral cutaneous femoral nerve. There are studies in the literature reporting that it provides effective analgesia after hip surgery.

Pericapsular nerve group block (PENG block) is a novel fascial block defined by Arango et al. In this block, it is aimed to block the femoral nerve and the accessory obturatory nerve by injecting local anesthetic between the pubic ramus and the psoas tendon. By blocking these nerves, anterior hip analgesia is provided. It is a safe and effective method as it is applied superficially and under ultrasound guidance. In radiological and cadaver studies, it has been reported that total hip analgesia can be provided by blocking the lateral femoral cutaneous, genitofemoral, obturator, and femoral nerves when high volume is applied. Studies evaluating PENG block efficacy are limited in the literature. There is a study comparing PENG block and femoral nerve block, but there is no study comparing it with FICB yet.

This prospective, multicenter study aimed to compare the efficacy of PENG block and FICB for postoperative analgesia management in patients undergoing hip arthroplasty with a prosthesis. Our primary aim is to compare global recovery scores, and our secondary aim is to evaluate postoperative opioid consumption, pain scores (Numerical Rating Scale-NRS), and side effects (allergic reaction, nausea, vomiting, etc.) related with opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III, aged 50-80 years, who were scheduled for hip arthroplasty under general anesthesia, will be included in the study.

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* patients who do not accept the procedure

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | Change from baseline scores at postoperative 1, 2, 4, 8, 16, and 24 hours
  This scoring system includes evaluating emotional state (12 questions), physical comfort (12 questions), psychological support (7 questions), physical independence (12 questions), and pain (7 questions).

SECONDARY OUTCOMES:
Pain scores (Numerical Rating Scale-NRS) | Postoperative 1, 2, 4, 8, 16, and 24 hours
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores will be recorded at postoperative 1, 2, 4, 8, 16 and 24 hours
Opioid consumption | Postoperative 1, 2, 4, 8, 16, and 24 hours
  If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University Hospital, Istanbul, Bagcilar
  - Mugla Sıtkı Kocman University Hospital, Muğla

IPD SHARING:
Plan to Share IPD: No
The investigator's will not share IPD

REFERENCES:
- [Background] O'Reilly N, Desmet M, Kearns R. Fascia iliaca compartment block. BJA Educ. 2019 Jun;19(6):191-197. doi: 10.1016/j.bjae.2019.03.001. Epub 2019 Apr 24. No abstract available. PMID 33456890
- [Background] Pepe J, Ausman C, Tafti D, Madhani NB. Ultrasound-Guided Fascia Iliaca Compartment Block. 2025 Sep 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK518973/ PMID 30085515
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Ciftci B, Ahiskalioglu A, Altintas HM, Tekin B, Sakul BU, Alici HA. A possible mechanism of motor blockade of high volume pericapsular nerve group (PENG) block: A cadaveric study. J Clin Anesth. 2021 Nov;74:110407. doi: 10.1016/j.jclinane.2021.110407. Epub 2021 Jun 24. No abstract available. PMID 34175637